CLINICAL TRIAL: NCT01399944
Title: The Molecular Basis for a Broad Range of Phenotypes Related to hTAS2R38
Status: Completed | Type: Observational
Sponsor: Monell Chemical Senses Center (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Julie A. Mennella, Member, Monell Chemical Senses Center
Other Study IDs: 813211; F32DC011975-01A1 (NIH); R01DC011287-01 (NIH)
Record Dates: First submitted 2011-07-20; First posted 2011-07-22 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Healthy
Keywords: bitter taste; psychophysics; genetics; epigenetics; bitterness sensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva and taste tissue will be collected from individuals enrolled in the study.
Oversight: Data Monitoring Committee: No

SUMMARY:
This single-site, within-subject, experimental study is designed to test the hypothesis that individuals express taste receptors differently and have different sensitivities to bitter taste samples, which results from uneven expression. Subjects will include 100 racially and ethnically diverse, healthy adults. All subjects will provide saliva samples for genetic analysis and undergo taste testing with common psychophysical stimuli. From the pool of 100 subjects, 36 subjects from the common heterozygous group (PAV/AVI) and two from each homozygous group (AVI/AVI, nontaster and PAV/PAV, taster) will be invited to return for two additional sessions. During both sessions the investigators will 1) measure bitterness thresholds for PROP, a common psychophysical stimulus; 2) measure bitterness perception of several vegetables; 3) obtain a saliva sample and 4) collect taste papillae. The investigators will then isolate DNA and RNA from the taste papillae and isolate DNA from saliva to evaluate molecular differences over time and between individuals and how it relates to taste psychophysics. All psychophysical and cellular measurements will be done during both sessions so that the investigators can determine how much variation is observed over a one-week time period in both cellular phenotype and psychophysical phenotype.

ELIGIBILITY:
Inclusion Criteria:

* Key inclusion criteria include age 18-40 years; English speaking, and good health at the time of study participation.

Exclusion Criteria:

* Key exclusion criteria include cigarette smoking, which alters taste perception, oral disease and subjects undergoing Coumadin therapy. Subjects showing signs of oral disease, including tongue lesions or xerostomia will be excluded from tongue biopsy and therefore excluded from the study. Subjects undergoing Coumadin therapy will be excluded from tongue biopsy due to the risk of bleeding, and therefore excluded from the study. Subjects will not be excluded because of economic status, gender, race or ethnicity.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adults of all races and both genders (N=100) will be involved in the proposed research. Typically, our population of subjects is approximately 45% African American, 45% Caucasian, 6% Hispanic, and 4% Asian. This increased representation of under-represented minorities in our subject populations is reflective of the greater Philadelphia region and has been achieved, in part, through our outreach efforts advertising in local newspapers throughout the city.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2011-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Bitter taste thresholds | 2 days of testing (2 hours each)
  Thresholds for propylthiouracil (PROP) will be measured using modified Harris-Kalmus recognition thresholds.
Taste intensity and hedonic ratings of vegetables | 3 days of testing (1-2 hours each)
  Subjects will rate the intensity of five basic taste qualities (bitter, salt, sweet, sour, umami) and the liking of PROP, urea, quinine, caffeine, denatonium solutions and pureed vegetables using the general labelled magnitude scale (gLMS)
TAS2R Genotype | 1 day of testing (1-1.5 hours)
  Genotype of several TAS2Rs will be determined from DNA extracted from a saliva sample.
mRNA expression levels | 2 days of testing (2 hours each)
  Expression of taste and related genes will be determined from mRNA extracted from human taste tissue obtained via tongue biopsy.

SECONDARY OUTCOMES:
Dietary habits | 2 days (2 hours each)
  Subjects will complete a 24 hour diet recall on 2 days of testing.
biometrics | 1 day (1-1.5 hours)
  Height, weight, blood pressure and bioimpedance measurements will be taken.

CONTACTS AND LOCATIONS:
Overall Officials: Julie A. Mennella, PhD, Principal Investigator — Monell Chemical Senses Center
Locations (1):
- Monell Chemical Senses Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Lipchock SV, Mennella JA, Spielman AI, Reed DR. Human bitter perception correlates with bitter receptor messenger RNA expression in taste cells. Am J Clin Nutr. 2013 Oct;98(4):1136-43. doi: 10.3945/ajcn.113.066688. Epub 2013 Sep 11. PMID 24025627